CLINICAL TRIAL: NCT00225589
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Parallel Group Phase III Study Measuring Effects on Intima Media Thickness: an Evaluation Of Rosuvastatin 40 mg (METEOR)
Brief Title: A Study Measuring Effects on Intima Media Thickness: An Evaluation of Rosuvastatin 40 mg (METEOR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4522IL/0088; METEOR; D3562C00088 (Other: AstraZeneca)
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Hypercholesteremia
Keywords: Hypercholesteremia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin calcium
  Other Names: Crestor

SUMMARY:
The purpose of this trial is to see if rosuvastatin will be effective in decreasing the thickness of the walls of the arteries in the neck for people who already have some evidence of thickening of these walls.

ELIGIBILITY:
Inclusion Criteria:

* Maximum IMT >1.2 mm and 3.5 mm at any location in the carotid ultrasound studies conducted at both Visit 2 (Week -4) and Visit 3 (Week -2)
* Subjects with age and no other risk factor: Fasting LDL-C at Visit 1 (Week -6) is >120 mg/dL (3.1mmol/L) and <190 mg/dL (4.9 mmol/L)
* Subjects with 2 or more risk factors and a 10-year coronary heart disease (CHD) risk < 10%: Fasting LDL-C at Visit 1 (Week -6) is >120 mg/dL (3.1 mmol/L) and <160 mg/dL (4.1 mmol/L)

Exclusion Criteria:

* Use of pharmacologic lipid-lowering medications (eg, HMG-CoA reductase inhibitors, fibrate derivatives, bile acid binding resins, niacin or its analogues at doses >400 mg) within 12 months prior to Visit 1 (Week -6).
* Clinical evidence of coronary artery disease or any other atherosclerotic disease such as angina, MI, TIA, symptomatic carotid artery disease, CVA, CABG, PTCA, peripheral arterial disease, AAA.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840
Dates: Start 2002-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Assess the effects of rosuvastatin treatment on the change in the mean maximum intima media thickness (IMT) of the 12 vessel segments: the near & far walls of the CCA, the carotid bulb & the ICA

SECONDARY OUTCOMES:
Assess the effects of rosuvastatin treatment on the following variables, with the same analyses being applied to the IMT variables:
Change in the mean maximum IMT of the near & far walls of the right & left CCA, carotid bulb, ICA
Change in the mean IMT of the near & far walls of the right & left CCA
Change in LDL-C, TC, HDL-C, TG, nonHDL-C, ApoB, ApoA-I, nonHDL-C/HDL-C, & ApoB/ApoA-I
Change in inflammatory marker: C-reactive protein (CRP)
Safety & tolerability, by evaluating the incidence & severity of adverse events & abnormal laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Science Director, MD, Study Director — AstraZeneca
Locations (57):
- United States (20):
  - Research Site, Alhambra, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Brooklyn Center, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Glen Mills, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Kirkland, Washington
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Brussels (Anderlecht)
  - Research Site, Leuven
- Czechia (2):
  - Research Site, Prague
  - Research Site, Slaný
- Research Site, Kuopio, Finland
- France (21):
  - Research Site, Auboué
  - Research Site, Bagnolet
  - Research Site, Boulogne-Billancourt
  - Research Site, Briey
  - Research Site, Delme
  - Research Site, Drancy
  - Research Site, Fresnes-en-Woëvre
  - Research Site, Ivry-sur-Seine
  - Research Site, Jarny
  - Research Site, Les Lilas
  - Research Site, Marange-Silvange
  - Research Site, Mars-la-Tour
  - Research Site, Metz
  - Research Site, Meudon
  - Research Site, Montigny-lès-Metz
  - Research Site, Moûtiers
  - Research Site, Paris
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Thionville
  - Research Site, Yerres
  - Research Site, Yutz
- Germany (4):
  - Research Site, München, Bavaria
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Essen
  - Research Site, München
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
  - Research Site, Utrecht
- Norway (3):
  - Research Site, Bekkestua
  - Research Site, Oslo
  - Research Site, Skedsmokorset

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- [Derived] Peters SA, Bots ML, Lind L, Groenewegen KA, de Korte C, den Ruijter HM; METEOR study group. The impact of variability in ultrasound settings on the measured echolucency of the carotid intima-media. J Hypertens. 2013 Sep;31(9):1861-7. doi: 10.1097/HJH.0b013e3283623548. PMID 23868083
- [Derived] Lind L, Peters SA, den Ruijter HM, Palmer MK, Grobbee DE, Crouse JR 3rd, O'Leary DH, Evans GW, Raichlen JS, Bots ML; METEOR Study Group. Effect of rosuvastatin on the echolucency of the common carotid intima-media in low-risk individuals: the METEOR trial. J Am Soc Echocardiogr. 2012 Oct;25(10):1120-1127.e1. doi: 10.1016/j.echo.2012.07.004. Epub 2012 Aug 9. PMID 22884641
- [Derived] Peters SA, den Ruijter HM, Palmer MK, Grobbee DE, Crouse JR 3rd, O'Leary DH, Evans GW, Raichlen JS, Bots ML; METEOR Study Group. Biologically implausible carotid intima-media thickness measurement values: effects on rate of change over time. Curr Med Res Opin. 2012 Jun;28(6):891-9. doi: 10.1185/03007995.2012.689255. Epub 2012 Jun 6. PMID 22536884
- [Derived] Stein EA, Vidt DG, Shepherd J, Cain VA, Anzalone D, Cressman MD. Renal safety of intensive cholesterol-lowering treatment with rosuvastatin: a retrospective analysis of renal adverse events among 40,600 participants in the rosuvastatin clinical development program. Atherosclerosis. 2012 Apr;221(2):471-7. doi: 10.1016/j.atherosclerosis.2011.12.011. Epub 2012 Jan 3. PMID 22304793
- [Derived] Peters SA, den Ruijter HM, Palmer MK, Grobbee DE, Crouse JR 3rd, O'Leary DH, Evans GW, Raichlen JS, Lind L, Bots ML; METEOR Study Group. Manual or semi-automated edge detection of the maximal far wall common carotid intima-media thickness: a direct comparison. J Intern Med. 2012 Mar;271(3):247-56. doi: 10.1111/j.1365-2796.2011.02422.x. Epub 2011 Aug 11. PMID 21726301
- [Derived] Peters SA, Dogan S, Meijer R, Palmer MK, Grobbee DE, Crouse JR 3rd, O'Leary DH, Evans GW, Raichlen JS, Bots ML. The use of plaque score measurements to assess changes in atherosclerotic plaque burden induced by lipid-lowering therapy over time: the METEOR study. J Atheroscler Thromb. 2011;18(9):784-95. doi: 10.5551/jat.8169. Epub 2011 May 27. PMID 21617330
- [Derived] Peters SA, Palmer MK, Grobbee DE, Crouse JR 3rd, Evans GW, Raichlen JS, Bots ML; METEOR Study Group. Effect of number of ultrasound examinations on the assessment of carotid intima-media thickness changes over time: the example of the METEOR study. J Hypertens. 2011 Jun;29(6):1145-54. doi: 10.1097/HJH.0b013e328345d85e. PMID 21546878
- [Derived] Peters SA, Palmer MK, Grobbee DE, Crouse JR 3rd, O'Leary DH, Raichlen JS, Bots ML. C-reactive protein lowering with rosuvastatin in the METEOR study. J Intern Med. 2010 Aug;268(2):155-61. doi: 10.1111/j.1365-2796.2010.02230.x. Epub 2010 Mar 6. PMID 20412373
- [Derived] Bots ML, Palmer MK, Dogan S, Plantinga Y, Raichlen JS, Evans GW, O'Leary DH, Grobbee DE, Crouse JR 3rd; METEOR Study Group. Intensive lipid lowering may reduce progression of carotid atherosclerosis within 12 months of treatment: the METEOR study. J Intern Med. 2009 Jun;265(6):698-707. doi: 10.1111/j.1365-2796.2009.02073.x. Epub 2009 Mar 2. PMID 19298496
- [Derived] Crouse JR 3rd, Raichlen JS, Riley WA, Evans GW, Palmer MK, O'Leary DH, Grobbee DE, Bots ML; METEOR Study Group. Effect of rosuvastatin on progression of carotid intima-media thickness in low-risk individuals with subclinical atherosclerosis: the METEOR Trial. JAMA. 2007 Mar 28;297(12):1344-53. doi: 10.1001/jama.297.12.1344. Epub 2007 Mar 25. PMID 17384434
- [Derived] Crouse JR 3rd, Grobbee DE, O'Leary DH, Bots ML, Evans GW, Palmer MK, Riley WA, Raichlen JS; METEOR Study Group. Carotid intima-media thickness in low-risk individuals with asymptomatic atherosclerosis: baseline data from the METEOR study. Curr Med Res Opin. 2007 Mar;23(3):641-8. doi: 10.1185/030079907X178711. PMID 17355745